CLINICAL TRIAL: NCT05041218
Title: Gauging Active Modalities of Error Detection and Signaling Obtained by Neural Interfaces in the Cathlab: the GAME-ON Study
Brief Title: Neural Interfaces to Monitor Fatigue and Sleepiness in the Cathlab
Acronym: GAME-ON
Status: Completed | Type: Observational
Sponsor: University Hospital of Ferrara (Other)
Responsible Party: Principal Investigator, Gianluca Campo, Professor, University Hospital of Ferrara
Other Study IDs: OspFE_25082021
Record Dates: First submitted 2021-08-26; First posted 2021-09-10 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Coronary Artery Disease; Mental Stress; Stress, Psychological
Keywords: neural interfaces; attentional effort; mental fatigue; sleepiness; coronary artery disease; percutaneous coronary intervention
MeSH Terms: conditions — Coronary Artery Disease; Stress, Psychological; Mental Fatigue; Sleepiness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients undergoing coronary artery angiography and/or percutaneous coronary intervention: Consecutive patients with indication to perform coronary artery angiography and/or percutaneous coronary intervention at Ferrara University Hospital
  Interventions: Other: Neural Interfaces Electroencephalogram measurement on Operators

INTERVENTIONS:
Other: Neural Interfaces Electroencephalogram measurement on Operators — Electroencephalogram based neural interfaces acquired during the interventional procedure and during alpha attenuation protocols (AAP) and psychometric questionnaires. AAP and psychometrics are acquired at the beginning of the shift, before and after each procedure performed.

SUMMARY:
Improvement of patients' care and outcome is largely based on development and validation of drugs and technologies, especially in rapidly evolving fields as Interventional Cardiology. In fact, even though the optimal efficiency of a cathlab can be influenced by Interventional Cardiologist's mental workload, stress' accumulation and performance, little if any attention is paid to the monitoring and optimization of his/her mental status. Electroencephalogram (EEG)-based neural-interfaces are able to estimate workload, fatigue and the degree of sleepiness through spectral analysis techniques. In particular, the amplitude of alpha waves is a widely validated indicator of mental engagement's level.

Developing a low cost and highly feasible device to monitor and analyze operator's mental engagement level and performance could be extremely appealing, especially considering both the lack of data in literature for interventional disciplines and the recent technology developments.

DETAILED DESCRIPTION:
The investigators will prospectively record and analyze Electroencephalogram (EEG) signals from 5 interventional cardiologists and 2 fellows in training in all consecutive procedures at Ferrara University Hospital. Considering the hypothesis of independence of the working shifts, given the heterogeneity of their structure in terms of procedures' number and type and their distance in time, it is then possible to assume that the same operator's psycho-physical state diverges between two different acquisition days. Muse S (InteraXon; Canada), a minimally invasive device paired via Bluetooth to a dedicated app, is used to record EEG signals. Neurometrics will be acquired during Alpha Attenuation Protocols (AAP), a sensitive test to quantify sleepiness which involves measuring alpha power during 2 cycle of eye opening/closing protocol, for a total amount of 4 minutes. AAP will be recorded at the beginning of the shift, before and after each procedure performed and allow to extrapolate waves' power measures obtained during resting condition (AA Coefficient-eyes open (AAC-eo), AAC-eyes closed (AAC-ec) and AAC-mean), related to fatigue, and AAC-ec/AAC-eo (AAC-ratio), related to sleepiness. In addition, alpha-prevalence (AP) during on-task will be measured. Alpha prevalence is an estimate of alpha-power. Investigators will also measure several validated psychometric questionnaires: Karolinska Sleepiness Scale (KSS), Sleep Quality Scale (SQS) and Profile of Mood States-Fatigue subscale (POMS-F). Heart rate variability (HRV) during tasks, related to psycho-physical stress, is assessed through the square root of the mean of the sum of squares of differences between adjacent normal R-R (rMSSD).

The Game-on project aims to describe workload, mental fatigue and sleepiness through variation of psychometric and neurometric measurements during a work shift with the intent of establishing determinants of error and lengthening of procedural times.

ELIGIBILITY:
Inclusion Criteria:

* indication to coronary artery angiography and/or percutaneous coronary intervention

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: consecutive patients undergoing invasive coronary artery angiography and/or percutaneous coronary intervention at Ferrara University Hospital
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2023-05-09 (Actual); Primary Completion 2025-03-24 (Actual); Study Completion 2025-03-24 (Actual)

PRIMARY OUTCOMES:
Sleepiness Sensitivity KSS | pre-procedure
  Sensitivity: proportion of operators with positive AAC ratio (AAC ratio values above study population median value are considered associated with sleepiness) of positive KSS questionnaire ones (true positive). KSS is defined as positive for values above preliminary study population median value (two months sampling of the same population between February and March 2021).
Sleepiness Sensitivity SQS | pre-procedure
  Sensitivity: proportion of operators with positive AAC ratio of positive SQS questionnaire ones (true positive). SQS is defined as positive for values above preliminary study population median value (two months sampling of the same population between February and March 2021).
Sleepiness Specificity KSS | pre-procedure
  Specificity: proportion of operators with negative AAC ratio (AAC ratio values below study population median value are not considered associated with sleepiness) of negative KSS questionnaire ones (true negative). KSS is defined as negative for values below preliminary study population median value (two months sampling of the same population between February and March 2021).
Sleepiness Specificity SQS | pre-procedure
  Specificity: proportion of operators with negative AAC ratio (AAC ratio values below study population median value are not considered associated with sleepiness) of negative SQS questionnaire ones (true negative). SQS is defined as negative for values below preliminary study population median value (two months sampling of the same population between February and March 2021).
Fatigue Sensitivity POMS-F | pre-procedure
  Sensitivity: proportion of operators with positive AAC ec/eo/mean (AAC ec/eo/mean values above study population median value are considered associated with fatigue) of positive POMS-F questionnaire ones (true positive). POMS-F is defined as positive for values above preliminary study population median value (two months sampling of the same population between February and March 2021).
Fatigue Specificity POMS-F | pre-procedure
  Specificity: proportion of operators with negative AAC ec/eo/mean (AAC ec/eo/mean values below study population median value are not considered associated with fatigue) of negative POMS-F questionnaire ones (true negative). POMS-F is defined as negative for values below preliminary study population median value (two months sampling of the same population between February and March 2021).
On task psycho-physical stress NASA-TLX | intraprocedure
  Proportion of operators with positive Alpha Prevalence (AP) eo (AP eo values above study population median value are considered associated with psychophysical stress) at the beginning of the procedure, end of the procedure and mean value during the procedure of operators with positive NASA-Task Load Index (TLX) (NASA-TLX value above preliminary study population median value (two months sampling of the same population between February and March 2021)).
On task psycho-physical stress rMSSD | intraprocedure
  Proportion of operators with positive AP eo (AP eo values above study population median value are considered associated with psychophysical stress) at the beginning of the procedure, end of the procedure and mean value during the procedure of operators with positive rMSSD (rMSSD value below preliminary study individual's mean value).
Correlation AP and rMSSD | intraprocedure
  Evaluate the correlation between AP and rMSSD curve during the procedure. Curves are built by evaluating AP and rMSSD values in 5 minutes slots all along the procedure.

SECONDARY OUTCOMES:
AUC Fatigue POMS-F (positive) | pre-procedure
  Area under the curve (AUC) of AAC eo/ec/mean positive for POMS-F positive
AUC Sleepiness KSS/SQS | pre-procedure
  Area under the curve (AUC) of AAC ratio positive for KSS/SQS positive
Procedural lengthening | intraprocedure
  To discriminate whether positive AAC eo at the beginning of the procedure, at the end of the procedure and the mean value during the procedure is associated with longer procedure time, higher contrast volume and x-ray time after correction for confounders (clinical presentation, number of treated vessels, calcifications, etc.)

CONTACTS AND LOCATIONS:
Overall Officials: Simone Biscaglia, MD, Principal Investigator — Azienda Ospedaliero Universitaria di Ferrara; Gianluca Campo, MD, Study Chair — Azienda Ospedaliero Universitaria di Ferrara
Locations (1):
- University Hospital of Ferrara, Ferrara, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Puma S, Matton N, Paubel PV, Raufaste E, El-Yagoubi R. Using theta and alpha band power to assess cognitive workload in multitasking environments. Int J Psychophysiol. 2018 Jan;123:111-120. doi: 10.1016/j.ijpsycho.2017.10.004. Epub 2017 Oct 7. PMID 29017780
- [Background] Brouwer AM, Hogervorst MA, van Erp JB, Heffelaar T, Zimmerman PH, Oostenveld R. Estimating workload using EEG spectral power and ERPs in the n-back task. J Neural Eng. 2012 Aug;9(4):045008. doi: 10.1088/1741-2560/9/4/045008. Epub 2012 Jul 25. PMID 22832068
- [Background] Morales JM, Ruiz-Rabelo JF, Diaz-Piedra C, Di Stasi LL. Detecting Mental Workload in Surgical Teams Using a Wearable Single-Channel Electroencephalographic Device. J Surg Educ. 2019 Jul-Aug;76(4):1107-1115. doi: 10.1016/j.jsurg.2019.01.005. Epub 2019 Jan 26. PMID 30691989
- [Background] Putilov AA, Donskaya OG. Alpha attenuation soon after closing the eyes as an objective indicator of sleepiness. Clin Exp Pharmacol Physiol. 2014 Dec;41(12):956-64. doi: 10.1111/1440-1681.12311. PMID 25224885